CLINICAL TRIAL: NCT04905862
Title: Multi Center Study to Assess the Humoral and Cellular Response After Vaccination Against COVID-19 in Patients Treated With Renal Replacement Therapy
Brief Title: Assessment of Immune Response After Vaccination Against COVID-19 in Patients Treated With Renal Replacement Therapy
Acronym: COViNEPH-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Leszek Tylicki, Professor, Medical University of Gdansk
Other Study IDs: COViNEPH-1
Record Dates: First submitted 2021-05-27; First posted 2021-05-28 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2021-08

CONDITIONS: Kidney Failure, Chronic; Covid19; Vaccine Reaction; Vaccine Adverse Reaction
Keywords: COVID-19; Vaccine; Dialysis; Immunity; Kidney transplant recipient
MeSH Terms: conditions — Kidney Failure, Chronic; COVID-19 | interventions — Immunity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hemodialyzed patients: Hemodialyzed patients vaccinated with BNT162b2 - mRNA vaccine against COVID-19
  Interventions: Diagnostic Test: Immune response; Other: Solicited common and expected adverse reactions shortly following vaccination (reactogenicity), use of antipyretic or pain medications and unsolicited adverse events and serious adverse events
- Patients treated with peritoneal dialysis: Patients treated with peritoneal dialysis vaccinated with BNT162b2 - mRNA vaccine against COVID-19
  Interventions: Diagnostic Test: Immune response; Other: Solicited common and expected adverse reactions shortly following vaccination (reactogenicity), use of antipyretic or pain medications and unsolicited adverse events and serious adverse events
- Patients without chronic kidney disease: Patients without chronic kidney disease vaccinated with mRNA BNT162b2 - vaccine against COVID-19
  Interventions: Diagnostic Test: Immune response; Other: Solicited common and expected adverse reactions shortly following vaccination (reactogenicity), use of antipyretic or pain medications and unsolicited adverse events and serious adverse events
- Kidney transplant recipients: Kidney transplant recipients vaccinated with mRNA vaccine against COVID-19
  Interventions: Diagnostic Test: Immune response; Other: Solicited common and expected adverse reactions shortly following vaccination (reactogenicity), use of antipyretic or pain medications and unsolicited adverse events and serious adverse events

INTERVENTIONS:
Diagnostic Test: Immune response — 1. Venous blood samples will be collected at seven-time points: before dose 1 of vaccine, 21 days after dose 1, within 14-21 days after dose 2 and 3,6,9,12 months after vaccination. From the volume of about 8 ml of the patient's peripheral blood, a fraction of PBMC (peripheral blood mononuclear cells) will be isolated.
  2. The level of antibodies against the SARS-CoV-2 nucleocapsid (N) antigen will be detected in serum using the Abbot Architect™SARS-CoV-2 IgG test.
  3. The level of neutralizing IgG and IgA antibodies against the SARS-CoV (S1 and S2 subunits) (S) will be detected in serum using the DiaSorin LIAISON®SARS-CoV-2 S1/S2 IgG serology COVID-19 S-Protein (S1RBD) Human IgA ELISA Kit respectively.
  4. The cellular component of the immune response will be tested using the ELISPOT method, which involves testing the amount of INF-γ and IL-2 released from leukocyte cells.
Other: Solicited common and expected adverse reactions shortly following vaccination (reactogenicity), use of antipyretic or pain medications and unsolicited adverse events and serious adverse events — The grading scales for side effects used in this study will derive from the FDA Center for Biologics Evaluation and Research guidelines on toxicity grading scales for volunteers enrolled in preventive vaccine clinical trials. Solicited reactions will be obtained 7 days after the first and the second dose, and 30 days after the final vaccination. Unsolicited adverse events and serious adverse events will be observed recorded through 1 month after the second dose

SUMMARY:
Chronically dialyzed patients and kidney transplant recipients have been identified as particularly vulnerable to SARS-CoV-2 infection due to unavoidable exposure. They have also high rates of comorbid conditions and have varying degrees of immunosuppression, which puts them at risk of developing very severe forms of COVID-19 disease with fatality rates varying from 16% to 32%. In such circumstances vaccination is the only chance to improve their extremely poor prognosis. There is very little published data on the response to vaccination in dialyzed patients and kidney transplant recipients so far. No data are available on the efficacy of vaccines against COVID-19 in patients treated with peritoneal dialysis (PD). Furthermore, given the fact that disturbances of acquired immunity in dialyzed patients are many and diverse it is uncertain whether vaccinating against SARS CoV-2 in these population will result in sufficient immune response and, by consequence, protection against infection. Registration studies on the basis of which population vaccinations are actually conducted were performed only in the general population. There were no dialyzed patients and kidney transplant recipients in the study groups, so these patients are vaccinated with doses and schedules for people without chronic kidney disease. It is not known whether vaccination under such standard schedule produces a sufficient immune response in them and how long it lasts. That's why the aim of this study is to evaluate the humoral and cellular immune response after mRNA vaccine against COVID-19 with which patients treated with renal replacement therapy are vaccinated in Poland. It will be a prospective, observational controlled study conducted in patients treated with renal replacement therapy (hemodialyzed subjects, patients treated with peritoneal dialysis and kidney transplant recipients) vaccinated with mRNA vaccine against COVID-19 according to common rules and manufactures recommendations.The control group will be made up of sex and age matched people without chronic kidney disease.The first goal of the study is to analyze seroconversion rate and titer magnitude of neutralizing IgG and IgA antibodies directed against spike (s) SARS-CoV-2 antigen after the first and the second dose of mRNA vaccine as well as after 3, 6, 9, 12 months after vaccination. The second goal is to evaluate the cellular immune response tested using the ELISPOT method at the same time points as above.The immune response will be compared to patients without chronic kidney disease as well as between hemodialysis, peritoneal dialysis patients and kidney transplant recipients.

DETAILED DESCRIPTION:
1. Venous blood samples will be collected at seven-time points: before dose 1 of vaccine, 21 days after dose 1, within 14-21 days after dose 2 and 3,6,9,12 months after vaccination. From the volume of about 8 ml of the patient's peripheral blood, a fraction of PBMC (peripheral blood mononuclear cells) will be isolated, which in the first stage of the study will be frozen in nitrogen. To generate serum, blood samples were centrifuged at room temperature at 2500 RPM for 10 minutes, aliquoted, frozen in -70˚C, and stored until use.
2. The level of antibodies against the SARS-CoV-2 nucleocapsid (N) antigen will be detected in serum using the Abbot Architect™SARS-CoV-2 IgG test.
3. The level of neutralizing IgG and IgA antibodies against the SARS-CoV (S1 and S2 subunits) (S) will be detected in serum using the DiaSorin LIAISON®SARS-CoV-2 S1/S2 IgG serology COVID-19 S-Protein (S1RBD) Human IgA ELISA Kit respectively.
4. The cellular component of the immune response will be tested using the ELISPOT method, which involves testing the amount of INF-γ and IL-2 released from leukocyte cells.
5. The grading scales for side effects (the same as in the pivotal trial) used in this study were derived from the FDA Center for Biologics Evaluation and Research (CBER) guidelines on toxicity grading scales for healthy adult volunteers enrolled in preventive vaccine clinical trials.
6. All medical data of patients from all groups will be extracted from their medical records.

ELIGIBILITY:
Inclusion Criteria:

* patients on chronic dialysis (hemodialysis or peritoneal dialysis) for at least 1 months and had received vaccination with mRNA vaccine BNT162b2 (BionTech/Pfizer Comirnaty) with a 3-week interval between first and second doses.

Exclusion Criteria:

* (-)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in:
  1. Department of Nephrology Transplantology and Internal Medicine, Medical University of Gdansk.
  2. NZOZ Diaverum Hemodialysis Unit in Gdynia.
  3. The University Centre of Maritime and Tropical Medicine in Gdynia
  4. 7th Naval Hospital in Gdansk
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Humoral immune response | 12 months (7 time points)
  Neutralizing IgG antibodies against the SARS-CoV (S1 and S2 subunits) (S)
Humoral immune response | 12 months (7 time points)
  Neutralizing IgA antibodies against the SARS-CoV (S1 and S2 subunits) (S)
The cellular immune response. | 12 months (7 time points)
  Testing the amount of INF-γ and IL- 2 released from leukocyte cells in response to stimulation with S proteins

SECONDARY OUTCOMES:
Solicited and unsolicited local and systemic reactogenicity | Until 1 month after the second dose
  Solicited common and expected adverse reactions shortly following vaccination (reactogenicity), use of antipyretic or pain medications and unsolicited adverse events and serious adverse events, i.e. those reported by the participants without prompts from the medical staff or observed by their physicians through 1 month after the second dose.

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Medical University of Gdansk, Gdansk, Pomeranian Voivodeship
  - 7th Naval Hospital in Gdansk, Gdansk
  - NZOZ Diaverum Gdynia, Gdynia
  - The University Centre of Maritime and Tropical Medicine in Gdynia, Gdynia

REFERENCES:
- [Derived] Piotrowska M, Zielinski M, Tylicki L, Biedunkiewicz B, Kubanek A, Slizien Z, Polewska K, Tylicki P, Muchlado M, Sakowska J, Renke M, Sudol A, Dabrowska M, Lichodziejewska-Niemierko M, Smiatacz T, Debska-Slizien A, Trzonkowski P. Local and Systemic Immunity Are Impaired in End-Stage-Renal-Disease Patients Treated With Hemodialysis, Peritoneal Dialysis and Kidney Transplant Recipients Immunized With BNT162b2 Pfizer-BioNTech SARS-CoV-2 Vaccine. Front Immunol. 2022 Jul 22;13:832924. doi: 10.3389/fimmu.2022.832924. eCollection 2022. PMID 35935974